CLINICAL TRIAL: NCT03991546
Title: Quantifying Pain and Narcotic Usage Following Orthopedic Surgery Using a Text-Messaging Robot
Brief Title: Pain and Narcotic Usage After Orthopaedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Anthony (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor-Investigator, Christopher Anthony, Orthopaedic Surgery Graduate Medical Education Resident 5, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201412701
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Fractures, Closed; Pain, Postoperative; Pain Catastrophizing; Pain, Acute; Analgesia; Opioid Use; Acceptance and Commitment Therapy; Orthopedics; Analgesics, Opioid; Text Messaging
Keywords: Opioid Pain Medication; PROMIS
MeSH Terms: conditions — Fractures, Closed; Pain, Postoperative; Acute Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Two study groups. The intervention group and the control group that does not receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental): Subjects randomizing into this arm received the study intervention that consisted of twice-daily, AM and PM, text messages starting on postoperative day one and ending on postoperative day fourteen. Subjects were only required to read these messages, which utilized the principles of Acceptance and Commitment therapy.
  Interventions: Behavioral: Acceptance and Commitment Therapy Delivered via an Automated Mobile Messaging Robot
- Control group (No Intervention): Subjects randomizing into this arm did not receive the text message study intervention.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy Delivered via an Automated Mobile Messaging Robot — Mobile messages utilizing the principles of Acceptance and Commitment therapy. These messages were developed in collaboration with a pain psychologist who specializes in treating chronic pain with Acceptance and Commitment therapy. Subjects received twice-daily messages for two weeks following their orthopaedic procedure.
  Arms: Acceptance and Commitment Therapy

SUMMARY:
This study aims to 1) observe the course of pain, 2) utilization of opioid pain medication, and 3) possible effect of a behavioral intervention delivered via an automated mobile phone messaging robot in patients undergoing surgical treatment of a traumatic orthopaedic injury.

DETAILED DESCRIPTION:
Adult patients presenting to a University Hospital Level 1 trauma center indicated for operative fixation of a traumatic upper or lower fracture were considered for the study. A partial Health Insurance Portability and Accountability Act waiver was granted for this investigation to allow research team members to review potential subject's medical record for any condition meeting exclusion criteria. Eligible patients consenting to the study will be assigned a unique study identification number (ID). A master database linking patient ID to patient name and medical record number will be housed on a password protected and encrypted departmental server location, which only research personnel can access.

Participants will complete a basic demographics survey and preoperative/baseline patient reported outcome surveys at enrollment, including the Patient-reported outcomes measurement information system (PROMIS) Pain Intensity 1A short form, PROMIS Pain Intensity 3A short form, PROMIS Pain Interference 8A short form, and PROMIS 8A Emotional Distress-Anxiety 8A short forms. Following completion of these surveys, subjects will be randomized in a 1:1 ratio using a random number generator into one of two study groups. The intervention group will receive mobile messages communicating the behavior intervention following surgery. The control group will not receive the intervention. Subjects will not be blinded to their study group. Participants randomized to the intervention group were subsequently enrolled into the automated mobile messaging protocol and received a confirmation message welcoming them to the study, which was reviewed with them by the research assistant. Subjects were instructed that they were only required to read all messages, no responses were required. No other aspects of patient care including surgical approaches, medications prescribed, or postoperative instructions differ between groups.

After completion of enrollment and assignment of study group, each participant's medical record will be reviewed to obtain the following data that will be recorded in the research study database: Age, Sex, BMI, Medical Comorbidities, Psychological Comorbidities, Substance Abuse History, and presence of preoperative outpatient opioid pain medication utilization.

Subjects in the intervention group will being receiving the mobile messaging intervention the day following surgery. The mobile messaging intervention consists of twice per day mobile messages, morning and evening, starting on postoperative day one and ending on postoperative day 14. Messages communicated to study participants employ the principles of Acceptance and Commitment therapy, otherwise known as ACT, which has been used in the treatment of chronic pain. Prior to discharge, patients will be seen by a research team member to review the opioid pain medication they are prescribed at discharge and instructed to have their pill bottle available to them to provide a pill count at follow-up.

A single instance of follow-up will take place on postoperative day 14. This will occur either in clinic or over the phone with a research team member. At this time, participants will be asked how many tablets of their opioid pain medication they consumed since discharge and to confirm with the amount tablets remaining. Additionally, subjects will fill out a second set of the patient reported outcome surveys completed at enrollment. Collection of these follow-up items marks the end of the subject's participation in the study. No data collection planned following the two week study period.

The study hypothesis is that subjects receiving the behavior intervention delivered via an automated mobile messaging robot would report consuming less opioid pain medication during the study period, and demonstrate better patient reported outcome survey scores than controls at follow-up.

An initial pilot cohort was recruited in order to obtain the data to run the power analysis that determined the population size for the randomized portion of the study. The preliminary study recorded the amount of opioid medication tablets utilized by these patients over a two-week postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Must have their own personal phone capable of sending and receiving text messages
* Must be familiar with sending and receiving text messages
* Must have a traumatic upper or lower extremity fracture
* Must be indicated for primary operative fixation of their orthopaedic injury

Exclusion Criteria:

* Any open orthopaedic injuries
* Current or previous infection at the injury site
* Cause of injury is self inflicted non-accidental trauma
* Active diagnosis of a pain syndrome or chronic condition requiring long-term pain medication usage
* Indication for fracture temporization using external fixation.
* Indication for revision surgery for non-union or hardware failure
* Bilateral upper extremity injuries impeding patient's ability to use a mobile phone
* Orthopaedic injuries limited to the distal hand and/or foot
* Preoperative admission to an intensive care unit (ICU)
* Active cancer diagnosis or history of malignancy receiving treatment within the last 5 years
* Presence of altered mental status, intellectual disability, or dementia, which impedes a patient from ethically providing consent.
* Indication for primary arthroplasty treatment of the traumatic injury

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Number of opioid pain medication tablets consumed | Measurement of outcome obtained on postoperative day fourteen.
  Amount of outpatient opioid pain medication consumed by participating subjects during the study period. Recorded as tablets consumed allowing for the calculation of morphine milliequivalents. Collected via a pill count in clinic or over the phone.
Change in reported pain intensity score (PROMIS Pain Intensity 1A) | Measurements assessed in person via the standardized forms listed above on the day of surgery (enrollment) and on postoperative day fourteen, in clinic or via telephone.
  Patient-reported outcomes measurement information system Pain Intensity (PROMIS) 1A short form scores collected from all participating subjects.
  PROMIS Pain Intensity 1A short form is a 1 question survey measuring an individual's average pain over the past 7 days. It utilizes a scale of 0 (no pain) to 10 (worst imaginable pain). Higher values represent worse pain outcomes.
  More information on this instrument, including a scoring manual, can be found at http://www.healthmeasures.net.
Change in reported pain intensity score (PROMIS Pain Intensity 3A) | Measurements assessed in person via the standardized forms listed above on the day of surgery (enrollment) and on postoperative day fourteen, in clinic or via telephone.
  Patient-reported outcomes measurement information system Pain Intensity (PROMIS) 3A short form scores collected from all participating subjects.
  PROMIS Pain Intensity 3A short form is a 3 question survey measuring an individual's pain over the past 7 days. It utilizes a scale of 1 (no pain) to 5 (very severe pain) for all questions. The scores for the 3 questions are summed and then matched to a corresponding t-score for the instrument. The corresponding t-score is the final, reportable score and can range from 30.7 to 71.8 for the PROMIS Pain Intensity 3A instrument. Higher t-score values represent worse pain outcomes.
  More information on this instrument, including a scoring manual, can be found at http://www.healthmeasures.net.
Change in reported pain interference score | Measurements assessed in person via the standardized forms listed above on the day of surgery (enrollment) and on postoperative day fourteen, in clinic or via telephone.
  Patient-reported outcomes measurement information system (PROMIS) Pain Interference 8A short form scores collected from all participating subjects.
  The PROMIS Pain Interference 8A short form is an 8 question survey that measures how much pain has interfered in the respondent's life over the past 7 days. It utilizes a scale of 1 (not at all) to 5 (very much) for all questions. The scores for all 8 questions are summed and then matched to a corresponding t-score for the instrument. The corresponding t-score is the final, reportable score and can range from 40.7 to 77.0 for the PROMIS Pain Interference 8A instrument. Higher t-score values represent worse pain interference outcomes.
  More information on this instrument, including a scoring manual, can be found at http://www.healthmeasures.net.
Change in reported emotional distress (anxiety) score. | Measurements assessed in person via the standardized forms listed above on the day of surgery (enrollment) and on postoperative day fourteen, in clinic or via telephone.
  Patient-reported outcomes measurement information system (PROMIS) Emotional Distress-Anxiety 8A short form scores collected from all participating subjects.
  The PROMIS Emotional Distress-Anxiety 8A short form is an 8 statement survey that measures how much emotional distress, specifically due to anxiety, a respondent has experienced over the past 7 days. It utilizes a scale of 1 (never) to 5 (always) for all the statements. The scores for all 8 statements are summed and then matched to a corresponding t-score for the instrument. The corresponding t-score is the final, reportable score and can range from 37.1 to 83.1 for the PROMIS Emotional Distress-Anxiety 8A instrument. Higher t-score values represent worse anxiety caused emotional distress outcomes.
  More information on this instrument, including a scoring manual, can be found at http://www.healthmeasures.net.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Anthony, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones J Jr, Southerland W, Catalani B. The Importance of Optimizing Acute Pain in the Orthopedic Trauma Patient. Orthop Clin North Am. 2017 Oct;48(4):445-465. doi: 10.1016/j.ocl.2017.06.003. PMID 28870305
- [Background] Hughes LS, Clark J, Colclough JA, Dale E, McMillan D. Acceptance and Commitment Therapy (ACT) for Chronic Pain: A Systematic Review and Meta-Analyses. Clin J Pain. 2017 Jun;33(6):552-568. doi: 10.1097/AJP.0000000000000425. PMID 27479642
- [Background] Nicholls JL, Azam MA, Burns LC, Englesakis M, Sutherland AM, Weinrib AZ, Katz J, Clarke H. Psychological treatments for the management of postsurgical pain: a systematic review of randomized controlled trials. Patient Relat Outcome Meas. 2018 Jan 19;9:49-64. doi: 10.2147/PROM.S121251. eCollection 2018. PMID 29403322
- [Background] Hayes SC. Acceptance and Commitment Therapy, Relational Frame Theory, and the Third Wave of Behavioral and Cognitive Therapies - Republished Article. Behav Ther. 2016 Nov;47(6):869-885. doi: 10.1016/j.beth.2016.11.006. Epub 2016 Nov 10. PMID 27993338
- [Background] Dindo L, Zimmerman MB, Hadlandsmyth K, StMarie B, Embree J, Marchman J, Tripp-Reimer T, Rakel B. Acceptance and Commitment Therapy for Prevention of Chronic Postsurgical Pain and Opioid Use in At-Risk Veterans: A Pilot Randomized Controlled Study. J Pain. 2018 Oct;19(10):1211-1221. doi: 10.1016/j.jpain.2018.04.016. Epub 2018 May 17. PMID 29777950
- [Background] Rathbone AL, Prescott J. The Use of Mobile Apps and SMS Messaging as Physical and Mental Health Interventions: Systematic Review. J Med Internet Res. 2017 Aug 24;19(8):e295. doi: 10.2196/jmir.7740. PMID 28838887
- [Background] Tofte JN, Anthony CA, Polgreen PM, Buckwalter JA, Caldwell LS, Fowler TP, Ebinger T, Hanley JM, Dowdle SB, Holte AJ, Arpey NC, Lawler EA. Postoperative care via smartphone following carpal tunnel release. J Telemed Telecare. 2020 May;26(4):223-231. doi: 10.1177/1357633X18807606. Epub 2018 Nov 14. PMID 30428766
- [Background] Anthony CA, Volkmar AJ, Shah AS, Willey M, Karam M, Marsh JL. Communication with Orthopedic Trauma Patients via an Automated Mobile Phone Messaging Robot. Telemed J E Health. 2018 Jul;24(7):504-509. doi: 10.1089/tmj.2017.0188. Epub 2017 Dec 20. PMID 29261036
- [Background] Anthony CA, Lawler EA, Glass NA, McDonald K, Shah AS. Delivery of Patient-Reported Outcome Instruments by Automated Mobile Phone Text Messaging. Hand (N Y). 2017 Nov;12(6):614-621. doi: 10.1177/1558944716672201. Epub 2016 Oct 6. PMID 29091492
- [Background] Day MA, Anthony CA, Bedard NA, Glass NA, Clark CR, Callaghan JJ, Noiseux NO. Increasing Perioperative Communication With Automated Mobile Phone Messaging in Total Joint Arthroplasty. J Arthroplasty. 2018 Jan;33(1):19-24. doi: 10.1016/j.arth.2017.08.046. Epub 2017 Sep 19. PMID 29017803
- [Background] Anthony CA, Lawler EA, Ward CM, Lin IC, Shah AS. Use of an Automated Mobile Phone Messaging Robot in Postoperative Patient Monitoring. Telemed J E Health. 2018 Jan;24(1):61-66. doi: 10.1089/tmj.2017.0055. Epub 2017 Jun 16. PMID 28622079
- [Background] Anthony CA, Polgreen LA, Chounramany J, Foster ED, Goerdt CJ, Miller ML, Suneja M, Segre AM, Carter BL, Polgreen PM. Outpatient blood pressure monitoring using bi-directional text messaging. J Am Soc Hypertens. 2015 May;9(5):375-81. doi: 10.1016/j.jash.2015.01.008. Epub 2015 Jan 21. PMID 25771023
- [Background] Anthony CA, Peterson AR. Utilization of a text-messaging robot to assess intraday variation in concussion symptom severity scores. Clin J Sport Med. 2015 Mar;25(2):149-52. doi: 10.1097/JSM.0000000000000115. PMID 24905538
- [Derived] Anthony CA, Rojas EO, Keffala V, Glass NA, Shah AS, Miller BJ, Hogue M, Willey MC, Karam M, Marsh JL. Acceptance and Commitment Therapy Delivered via a Mobile Phone Messaging Robot to Decrease Postoperative Opioid Use in Patients With Orthopedic Trauma: Randomized Controlled Trial. J Med Internet Res. 2020 Jul 29;22(7):e17750. doi: 10.2196/17750. PMID 32723723